CLINICAL TRIAL: NCT04920656
Title: Universal Genetic Testing Versus Guidelines-Directed Testing for Germline Pathogenic Variants Among Non-Western Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Principal Investigator, Hikmat Abdel-Razeq, Professor, Chairman of department of medicine, Chief Medical officer, Deputy Director General, King Hussein Cancer Center
Other Study IDs: 20 KHCC 202
Record Dates: First submitted 2021-05-16; First posted 2021-06-10 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Breast cancer patients: All adult patients with a confirmed diagnosis of breast cancer, aged 18 or older at time of cancer diagnosis, will be invited to participate.

SUMMARY:
The study aims to examinethe pattern and frequency of pathogenic variants among all newly diagnosed breast cancer patients in a genetically distinct population. Additionally, the uptake rate of "cascade family screening" , frequency of pathogenic variants and barriers against testing will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, age ≥ 18 years at time of cancer diagnosis
* Pathology proven diagnosis of breast cancer (including DCIS); any stage. (prior history of cancer is allowed)
* Willingness to participate
* Signed consent form.

Exclusion Criteria:

- Major psychiatric disorder (defined as: patients followed by a psychiatrist and on antipsychotic medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who fulfill the inclusion/exclusion criteria, and are treated and followed up at KHCC will be invited.
  A total of 1000 patients are estimated to participate
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of pathogenic or likely pathogenic germline variants among newly diagnosed breast cancer patients tested by universal multigene panel testing or guideline-based targeted testing | 2021-2023
Number of participants with variants of uncertain significance (VUS) as assessed by universal multigene panel testing versus guideline-based targeted testing | 2021-2023
The reasons/ Barriers for refusal of genetic cascade testing among newly diagnosed cancer patients | 2021-2023

SECONDARY OUTCOMES:
Rate of cascade testing of family members of the participants with positive pathogenic mutation | 2021-2023
  The family of the positive patients will be offered the genetic testing.
Prevalence of pathogenic or likely pathogenic mutations among family members of the patients with pathogenic mutations using the universal multigene panel | 2021-2023
Prevalence of variants of uncertain significance (VUS) among tested family members of participants with pathogenic mutations as assessed by universal multigene panel testing | 2021-2023
The reasons/ Barriers for refusal of genetic cascade testing among family members of the tested patients with pathogenic mutations | 2021-2023

CONTACTS AND LOCATIONS:
Overall Officials: Hikmat Abdel-Razeq, Principal Investigator — King Hussein Cancer Center
Locations (1):
- King Hussein Cancer Center, Amman, Amman Governorate, Jordan